CLINICAL TRIAL: NCT01659866
Title: Evaluation of Directed Antimicrobial Prophylaxis for Transrectal Ultrasound Guided Prostate Biopsy (TRUSP)
Brief Title: Antibiotic Prophylaxis for Transrectal Prostate Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Anthony Schaeffer, Herman L. Kretschmer Professor and Chair, Department of Urology, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00059558; EAM-237 (Other: Excellence in Academic Medicine)
Record Dates: First submitted 2012-07-09; First posted 2012-08-08 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2016-09

CONDITIONS: Infection
Keywords: Infection; Antibiotic resistance; Prostate biopsy
MeSH Terms: conditions — Infections | interventions — Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Cefuroxime; Ceftriaxone; Gentamicins; Amikacin; Aztreonam; Imipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cipro-susceptible (Other): Patients with ciprofloxacin-susceptible bacteria on their rectal swab cultures will receive ciprofloxacin, the standard of care, as prophylaxis for their prostate biopsy
  Interventions: Drug: Ciprofloxacin
- Cipro-resistant (Active Comparator): Patients with ciprofloxacin-resistant bacteria on their rectal swab will receive one of the following drugs:
  * trimethoprim-sulfamethoxazole 1 double strength tablet orally 2 hours before the procedure and again 12 hours later
  * cefuroxime 500 mg orally 2 hours before the procedure then again 12 hours later
  * ceftriaxone 500 mg intramuscularly 2 hours before the procedure
  * gentamicin 2mg/kg intramuscularly 2 hours before the procedure
  * amikacin 5 mg/kg intramuscularly 2 hours before the procedure
  * aztreonam 500 mg intramuscularly 2 hours before the procedure
  * imipenem 500 mg intramuscularly 2 hours before the procedure
  * ceftriaxone 2000 mg intravenously 1 hour before the procedure
  * gentamicin 2 mg/kg intravenously 1 hour before the procedure
  * amikacin 5mg/kg intravenously 1 hour before the procedure
  * aztreonam 2000 mg intravenously 1 hour before the procedure
  * imipenem 1000 mg intravenously 1 hour before the procedure
  Interventions: Drug: trimethoprim-sulfamethoxazole; Drug: cefuroxime; Drug: ceftriaxone; Drug: gentamicin; Drug: amikacin; Drug: aztreonam; Drug: imipenem

INTERVENTIONS:
Drug: Ciprofloxacin — 500 mg orally 2 hours before prostate biopsy
  Arms: Cipro-susceptible
Drug: trimethoprim-sulfamethoxazole — 1 double strength tablet orally 2 hours before the procedure and again 12 hours later
  Arms: Cipro-resistant
Drug: cefuroxime — 500 mg orally 2 hours before the procedure then again 12 hours later
  Arms: Cipro-resistant
Drug: ceftriaxone — 500 mg intramuscularly 2 hours before the procedure
  Arms: Cipro-resistant
Drug: gentamicin — 2 mg/kg intramuscularly 2 hours before the procedure
  Arms: Cipro-resistant
Drug: amikacin — 5 mg/kg intramuscularly 2 hours before the procedure
  Arms: Cipro-resistant
Drug: aztreonam — 500 mg intramuscularly 2 hours before the procedure
  Arms: Cipro-resistant
Drug: imipenem — 500 mg intramuscularly 2 hours before the procedure
  Arms: Cipro-resistant
Drug: ceftriaxone — 2000 mg intravenously 1 hour before the procedure
  Arms: Cipro-resistant
Drug: gentamicin — 2 mg/kg intravenously 1 hour before the procedure
  Arms: Cipro-resistant
Drug: amikacin — 5 mg/kg intravenously 1 hour before the procedure
  Arms: Cipro-resistant
Drug: aztreonam — 2000 mg intravenously 1 hour before the procedure
  Arms: Cipro-resistant
Drug: imipenem — 1000 mg intravenously 1 hour before the procedure
  Arms: Cipro-resistant

SUMMARY:
This study is being conducted in men scheduled to undergo transrectal ultrasound-guided prostate biopsy (TRUSP). Traditionally prior to prostate biopsy, an antibiotic, ciprofloxacin, has been given to men to prevent biopsy-related infections. In recent years as ciprofloxacin resistance has increased in the community, more and more men are becoming infected with ciprofloxacin-resistant bacteria after prostate biopsy. This study is being done to determine if obtaining rectal swab cultures and choosing antibiotics based on these culture results will result in fewer infectious complications than giving all men ciprofloxacin.

The investigators will compare 2 groups: men whose rectal swabs do not show ciprofloxacin-resistant bacteria will receive ciprofloxacin prior to biopsy, and men whose swabs do show ciprofloxacin-resistant bacteria will receive alternative antibiotics based on their culture results. Our hypothesis is that these 2 groups will have equal numbers of post-biopsy infectious complications and both groups will have fewer infectious complications than a historical group who received empiric ciprofloxacin without the benefit of rectal swab culture results.

DETAILED DESCRIPTION:
This study is a prospective, nonrandomized trial evaluating the efficacy of directed antimicrobial prophylaxis prior to transrectal ultrasound-guided prostate biopsy (TRUSP) compared with ciprofloxacin prophylaxis, the current standard of care. Northwestern University will be the lead site. After signing informed consent, study participants will complete a pre-biopsy questionnaire to record demographics and assess for known risk factors for infection and will have a rectal swab obtained. Patients whose swabs indicate colonization with ciprofloxacin-susceptible gram-negative bacteria (CS-GNB) will receive ciprofloxacin as pre-procedure prophylaxis and those whose swabs indicate colonization with ciprofloxacin-resistant gram-negative bacteria (CR-GNB) will receive pre-procedure antimicrobial prophylaxis based on study protocol.

All patients will be contacted by phone twice after their biopsies, at approximately 7 and 30 days, to detail post-procedure infectious complications including fever, urinary tract infection, bacteremia and sepsis. Subjects who experience infections will have additional information regarding the infectious complications and cost of therapy abstracted from their medical record. The TRUSP results will also be recorded. Bacterial isolates from the rectal swabs will be archived.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* All individuals who will undergo TRUSP as part of their standard of care are eligible for study.

Exclusion Criteria:

* Men under 30 years of age
* Individuals whose rectal swab indicates that they harbor CS-GNB who cannot receive ciprofloxacin as pre-procedure prophylaxis for any reason
* Individuals whose rectal swab indicates that they harbor CR-GNB who cannot abide by the antimicrobial prophylaxis guidelines outlined in the study protocol for any reason
* Individuals who do not wish to complete the pre-procedure risk factor questionnaire or the two post-procedure phone questionnaires to assess for infectious complications

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Schaeffer, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Urology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zembower TR, Maxwell KM, Nadler RB, Cashy J, Scheetz MH, Qi C, Schaeffer AJ. Evaluation of targeted antimicrobial prophylaxis for transrectal ultrasound guided prostate biopsy: a prospective cohort trial. BMC Infect Dis. 2017 Jun 7;17(1):401. doi: 10.1186/s12879-017-2470-1. PMID 28592230

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 563 patients consented and of these, 53 were excluded as follows: 16 patients had issues with informed consent, 20 received antimicrobials off protocol, 16 did not undergo TRUSP and 1 was lost to follow up. Thus 510 patients underwent swabs; 430 had CS isolates while 80 had CR isolates. All 510 patients completed the study.
Period: Overall Study
Arm/Group | Cipro-susceptible | Cipro-resistant
Started | 430 | 80
Completed | 430 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men >/= 18 scheduled for transrectal prostate biopsy who signed consent underwent a rectal swab culture to determine whether they harbored ciprofloxacin-susceptible or -resistant flora. Antimicrobial prophylaxis was chosen based on this result, and patients were followed for 30 days to see if they developed an infection post-procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cipro-susceptible | Cipro-resistant | Total
Number analyzed (Participants) | 430 | 80 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.1) | 61.6 (7.6) | 62.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 430 | 80 | 510
Region of Enrollment [Number; unit: participants]
  United States | 430 | 80 | 510

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-biopsy Infection.
Description: To measure and compare the rates of infection following TRUSP in subjects with and without CR-GNB. This measure is number of participants with post-biopsy infection.
Time Frame: 30 days post-biopsy
Population: Of the 563 patients who signed consent, 53 were excluded; thus, 510 patients participated in the study. Of these 510, 430 harbored ciprofloxacin-susceptible flora and 80 harbored ciprofloxacin-resistant flora.
Measure: Number; unit: participants
Arm/Group | Cipro-susceptible | Cipro-resistant
Number analyzed (Participants) | 430 | 80
participants | 6 | 3
Statistical Analysis 1: Comparison: Cipro-susceptible vs Cipro-resistant; Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cipro-susceptible | Cipro-resistant
All-Cause Mortality (participants affected / at risk) | 0/430 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/430 | 0/80
Other Adverse Events (participants affected / at risk) | 0/430 | 0/80

LIMITATIONS AND CAVEATS:
Did not reach recruiting targets due to fewer prostate biopsies being performed than originally estimated in the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No